CLINICAL TRIAL: NCT06395064
Title: The Effect of Dimenhydrinate on Postoperative Nausea and Vomiting After Abdominal Hysterectomy: Randomized-controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Preeyaporn Jirakittidul (Other)
Responsible Party: Sponsor-Investigator, Preeyaporn Jirakittidul, Assist Prof Dr. Preeyaporn Jirakittidul, Mahidol University
Organization: Mahidol University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 313/2024
Record Dates: First submitted 2024-04-29; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Gynecologic Neoplasm; Healthy Women
Keywords: post-operative nausea vomiting
MeSH Terms: conditions — Genital Neoplasms, Female | interventions — Dimenhydrinate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dimenhydrinate (Active Comparator): Dimenhydrinate 50 mg
  Interventions: Drug: Dimenhydrinate
- Placebo (Placebo Comparator): NSS 10 ml
  Interventions: Drug: Dimenhydrinate

INTERVENTIONS:
Drug: Dimenhydrinate — Dimenhydrinate 50mg intravenously

SUMMARY:
The aim of this clinical trial is to learn if Dimenhydrinate works to prevent postoperative nausea-vomiting in adult women who undergoing abdominal hysterectomy. The primary question is: Does Dimenhydrinate lower the proportion of postoperative nauseavomiting during the day 1 after surgery. Researcher will compare Dimenhydrinate to a placebo (a-look-alike substance that contains no drug) which will give intravenously when the patient come back to the ward, to see if Dimenhydrinate work to prevent nauseavomiting during the postoperative day1. All participants will receive standard treatment during pre-operative, intra-operative and the immediate post-operative periods. Participants will receive Dimenhydrinate or placebo only one dose after discharge from the recovery room. During the day 1 postoperative, participants will report their symptoms and keep a diary of the number of tmes they use additional anti-emetic drugs.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years female
* undergoing trans abdominal hysterectomy

Exclusion Criteria:

* undergoing emergency surgery
* pregnancy or breastfed women
* post delivery less than 6 weeks
* history of allergic reaction or precaution to use the protocol drug
* BMI less than 18 or more than 30 kg/m2
* Need ICU care after surgery

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
occurrence and times of nausea vomiting | at ward, 6, 12, 24 hr postoperation

IPD SHARING:
Plan to Share IPD: No